CLINICAL TRIAL: NCT03144609
Title: Impact of Protective Mechanical Ventilation of Obese Patients on the Postoperative Respiratory Function During Oral Surgical Procedures
Brief Title: Mechanical Ventilation of Obese Patients During Oral Surgical Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klarić, Vlasta, M.D. (Individual)
Responsible Party: Principal Investigator, Klarić, Vlasta, M.D., Principal Investigator, Klarić, Vlasta, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vllastica
Record Dates: First submitted 2017-04-27; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: mechanical ventilation, obesity, oral-surgical procedures
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEEP 4 (Active Comparator): Active Comparator low PEEP: obese patient during oral-surgical procedures under general anesthesia ventilated with Positive endexpiratory pressure (PEEP) 4 cm H2O(water)
  Interventions: Procedure: low PEEP
- PEEP 7 & ARM (Experimental): Experimental ARM & Experimental high PEEP: obese patient during oral-surgical procedures under general anesthesia ventilated with PEEP( positive endexpiratory pressure) 7 cm H2O with ARM(alveolar recruitment maneuver) provided every 30 min
  Interventions: Procedure: ARM; Procedure: high PEEP
- PEEP 10 & ARM (Experimental): Experimental ARM & Experimental high PEEP:obese patient during oral-surgical procedures under general anesthesia ventilated with PEEP( positive endexpiratory pressure) 10 cm H2O with ARM(alveolar recruitment maneuver) provided every 30 min
  Interventions: Procedure: ARM; Procedure: high PEEP

INTERVENTIONS:
Procedure: low PEEP — The control group consisted of obese patients mechanically ventilated by a standardized volume-controlled breathing mode with low respiratory volume without alveolar recruitment maneuver and using low values of PEEP up to 4 cm H2O.
  Other Names: low positive endexpiratory pressure
  Arms: PEEP 4
Procedure: ARM — The experimental groups also consisted of obese patients mechanically ventilated by a volume-controlled breathing mode with low respiratory volume 7 ml/kg ideal body mass, but with alveolar recruitment maneuver performed immediately after induction, followed every 30 minutes during the hemodynamic stable condition under operation.
  Other Names: alveolar recruitment maneuver
  Arms: PEEP 10 & ARM; PEEP 7 & ARM
Procedure: high PEEP — The experimental groups also consisted of obese patients mechanically ventilated by a volume-controlled breathing mode with low respiratory volume 7 ml/kg ideal body mass, but with higher PEEP, provided that the upper limit of 40 cm H20 was not exceeded.
  Other Names: high positive endexpiratory pressure
  Arms: PEEP 10 & ARM; PEEP 7 & ARM

SUMMARY:
The prevalence of obese patients in a great number of patients scheduled for elective surgery under general anesthesia has been on the increase. Recent studies suggest an intraoperative protective mechanical ventilation for the obese. Surgical procedures in the oral cavity increase the risk of perioperative complications of obese patients. By making this randomized clinical study, investigators want to determine whether the protective intraoperative ventilation with the use of higher positive end-expiratory pressure and recruitment maneuvers compared to ventilation with low positive end-expiratory pressure and without recruitments cause better postoperative respiratory function parameters of obese patients during oral surgical procedures. Investigators also aim to establish the fact which value of a positive end-expiratory pressure has a favorable impact on the respiratory function without negative hemodynamic effect.

DETAILED DESCRIPTION:
Oral surgeries of obese patients in general endotracheal anesthesia are a special challenge as in the most extensive types of interventions any form of regional anesthesia is inadequate, duration of surgery is short but requires deep level of anesthesia after which a quick awakening and most rapid release from hospital are expected, with a known high perioperative risk complications of obese patients.

Oral surgical procedures in the oral cavity due to possible postoperative upper airway oedema increase the risk of postoperative hypoxia in obese patients. Therefore, it is important to intraoperatively mechanically ventilate obese patients with the aim of good ventilation-perfusion ratio without creating new atelectasis, to minimize the risk of postoperative respiratory decompensation and to provide rapid recovery.

As the prevalence of obesity in the world increases as chronic diseases, the number of obese patients scheduled for oral surgery is growing. Studies involving different ways of intraoperative mechanical ventilation of obese patients are mostly processed laparoscopic abdominal studies that can not exclude the additional effect of intraabdominal pressure on the formation of pulmonary atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* body mass index greater than 30 kg / m2
* surgical operation in the area of the oral cavity in general endotracheal anesthesia - cystectomy, alveotomy, mandible and maxilla osteosynthesis after jaw trauma, operation of retained and affected teeth, orthodontic surgical treatment of jaw deformity, benign tumor surgery
* ASA (American Society of Anesthesiologists) Classification of Patients 2-3
* duration of general endotracheal anesthesia from 1 to 2.5 hours

Exclusion Criteria:

* Allergy to anesthetics
* previous lung operations
* documented heart disease (NYHA II, III)
* Pulmonary disease (asthma, COPD)
* Obstructive pulmonary function disorders according to spirometry: FVC(forced vital capacity) may and may not be normal, FEV1(forced expiratory volume at one second) <80%, FEV1 / FVC <80%)
* neuromuscular disease
* clinical sign of cardiovascular disease established during preoperative treatment
* pregnancy
* Patients who, for some reason after surgery, have to remain intubated and mechanically ventilated in the Intensive Medicine Unit
* refuse to sign informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
preoperative and postoperative change in arterial blood gas analysis within and between groups of patients | Preoperative parameters were compared with change in early postoperative parameter. Early postoperative measurements were measurements after 15 minutes from the operation, then in the first and third hours, and 24 hours after the operation.
  preoperative blood gas analysis measured an hour before induction and compared with blood gas analysis measured four times in postoperative period, after three different strategies of mechanical ventilation.Blood gas analysis will be compared within a group and between the groups.

SECONDARY OUTCOMES:
change in preoperative and postoperative degree of dyspnoea measured on Visual Analog Scale | 25 perioperative hours.Preoperative degree was measured one hour before the start of the operation. Early postoperative measurements were measured 15 min after the operation started, then in the first, third and 24th hours after surgery
  the degree of dyspnea in the early postoperative period between and within groups and compared with preoperative status. The degree of dyspnoea was determined by the participants on the Visual Analog Scale (0-10). Change From Baseline in dyspnoea Scores on the Visual Analog Scale at 24 hours were measured.
The connection between the various risks of difficult intubation and obesity. | up to 1 day:Visual Scale Cormack- Lehane classification was measured at laryngoscopy for intubation by investigator, all other measurements were measured once at preoperative Anesthetic examination
  morphological characteristics of oral cavity of obese patients,as indicators of the risk of severe intubation, such as interdental spacing in open mouth, type of bite, Mallampati Classification , Cormack-Lehane classification, thyromental and sterno-mental distance and anatomical anomaly of the face . Compare their association with impaired ventilation and / or intubation according to body mass index through study completion
PEEP effects on MAP | 1-2,5 intraoperative hours.Intraoperative measurements were performed 5 min before and 5 min after induction, then every 30 minutes during operation.Change in MAP includes only period from the beginning operation to the end of surgery and extubation.
  intraoperative effect of different PEEP values on systemic circulatory stability by measuring systolic and diastolic blood pressure and mean arterial blood pressure (MAP).
ARM(alveolar recruitment maneuver) effects on MAP | 1-2,5 intraoperative hours.Intraoperative measurements were performed 5 min before and 5 min after induction, then every 30 min during operation, and 5 min after ARM is performed. Change in MAP includes period from the beginning to the end of operation
  intraoperative effect of lung recruitment maneuvers on systemic circulatory stability by measuring systolic and diastolic blood pressure and mean arterial blood pressure (MAP).

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Klarić, M.D., Principal Investigator

IPD SHARING:
Plan to Share IPD: No